CLINICAL TRIAL: NCT05483608
Title: Clinical Trial of Vertical Climbing Ergometer Exercise (CLMBR) in People With Chronic Low Back Pain
Brief Title: Vertical Climbing (CLMBR) Exercise for Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Jamie Mathew Wood, Program Manager, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 21-1568
Record Dates: First submitted 2022-07-31; First posted 2022-08-02 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Chronic Low Back Pain
Keywords: low back pain; exercise; vertical climbing
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The physician screening participants and the primary outcome assessor will be blinded to group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vertical climbing ergometer exercise (Experimental): 8 weeks of 3 times per week (24 sessions in total) of 30 minutes of vertical climbing ergometer exercise using the CLMBR. Intensity will be prescribed at a level of 12 to 14 on the Borg Rate of Perceived Exertion Scale.
  Interventions: Other: Vertical climbing ergometer exercise
- Recumbent cycling (Active Comparator): 8 weeks of 3 times per week (24 sessions in total) of 30 minutes of recumbent cycle ergometer exercise. Intensity will be prescribed at a level of 12 to 14 on the Borg Rate of Perceived Exertion Scale.
  Interventions: Other: Recumbent cycling

INTERVENTIONS:
Other: Vertical climbing ergometer exercise — Exercise using the CLMBR, a vertical climbing exercise ergometer.
  Arms: Vertical climbing ergometer exercise
Other: Recumbent cycling — Exercise using a recumbent cycle ergometer
  Arms: Recumbent cycling

SUMMARY:
This is a randomized control trial of vertical climbing ergometer exercise for individuals with chronic low back pain. Using a parallel-arm design, participants will be randomized to 8 weeks of supervised exercise using either the vertical climbing ergometer (CLMBR) or a recumbent cycling ergometer. This feasibility study will examine the safety, tolerability, and efficacy of vertical climbing exercise for individuals with chronic low back pain.

ELIGIBILITY:
Inclusion criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Confirmed chronic (>12 weeks) low back pain at screening assessment (based on patient history)
* Ability to comply with the current Mount Sinai Health system COVID-19 requirements for research participants (e.g., vaccination, masks)

Exclusion criteria:

* Criteria will be evaluated during the clinical evaluation at the screening visit. All determinations will be the decision of the study physician:
* Less than 2/10 low back pain on 0-10 numeric rating scale for average pain over past 7 days at baseline assessment
* Any cardiovascular or musculoskeletal contraindication to exercise
* Impaired balance contraindicating exercise
* Known psychological illnesses or cognitive impairments contraindicating exercise or preventing the ability to complete study assessments
* Current pregnancy
* Current medications or new medications commenced that may impact the ability for change to be detected in study
* Any other contraindication in the opinion of the study physician

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-11-12 (Actual); Study Completion 2023-11-12 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | 8 Weeks
  Incidence of adverse events
Number of completed exercise sessions | 8 Weeks
  The number of completed exercise sessions. A completed session is defined as achieving a minimum of 15 minutes of active exercise during a commenced session.
Change in Numeric Pain Rating Scale | Baseline and 8 Weeks
  11-point numerical rating scale evaluating average pain intensity over the past 7 days. A clinically meaningful difference will be considered as 2 points. Change in Numeric Pain Rating scale at 8 weeks as compared to baseline. Full scale from 0-10, with higher score indicating more pain.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale | 8 weeks
  Average acute change in pain intensity on 11-point numerical rating scale (higher = worse pain) during or immediately post-exercise, or reported at the beginning of the following session (unless believed that the change in pain was caused by something unrelated to the study intervention).
Minutes of exercise completed | 8 weeks
  Minutes of exercise completed during the exercise sessions.
Change in The Oswestry Disability Index | Baseline and 8 weeks
  The Oswestry Disability Index will be used to evaluate changes in disability in day-to-day activities as a result of low back pain. A clinically meaningful difference will be considered as 10 points. Full scale is 0 (no disability) to 50 (complete disability), higher score indicating poorer health outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Wood, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Union Square, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data will only be shared upon reasonable request